CLINICAL TRIAL: NCT01338363
Title: Drug Utilization and Safety Events Among Children Using Esomeprazole, Other Proton Pump Inhibitors or H2-receptor Antagonists
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: PHARMO Institute for Drug Outcome Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: D9612N00016
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Hospitalized Cases of Angioneurotic Oedema; Pneumonia; Gastroenteritis; Failure to Thrive; Seizures; Acute Interstitial Nephritis and Thrombocytopenia
Keywords: acid suppressing drugs; pharmacoepidemiology; children
MeSH Terms: conditions — Pneumonia; Gastroenteritis; Failure to Thrive; Seizures; Acute Tubulointerstitial Nephritis; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (3):
- All first time users of esomeprazole
- All first time users of other PPIs
- All first time users of H2-receptor antagonists

SUMMARY:
The purpose of this study is

1. To describe patient characteristics and drug usage among children that are prescribed esomeprazole for the first time and to compare them with patients who are prescribed other proton pump inhibitors (PPIs) or H2-receptor antagonists for the first time.
2. To ascertain all incident hospitalized cases of angioneurotic oedema, pneumonia, gastroenteritis, failure to thrive, convulsions/seizures, acute interstitial nephritis and thrombocytopenia among new users in the three cohorts of esomeprazole, other PPIs and H2-receptor antagonists.

DETAILED DESCRIPTION:
Time Perspective: Other = Retrospective analysis of prospectively collected data Number of Anticipated Subjects: All subjects dispensed esomeprazole, other PPIs or H2-receptor antagonists for the first time during the study period

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years
* Newly dispensed esomeprazole, other proton pump inhibitors or H2-receptor antagonists

Exclusion Criteria:

* Children with less than one year of history in PHARMO RLS before study cohort entry (if a child is <1 year at cohort entry, history from birth is required)
* Children using more than 1 acid suppressing drug concomitantly at cohort entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all children aged 0 to 18 years receiving a first dispension of acid suppressing drugs recorded in the PHARMO RLS database between September 2008 and October 2011. Subjects will be followed-up for at least 18 month. First review of study outcomes including chart reviews is estimated to start in August 2011.
Sampling Method: Non-Probability Sample
Enrollment: 23470 (Actual)
Dates: Start 2011-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Drug utilization: Description of patient characteristics and drug usage | Study period 3 years
Follow-up of safety outcomes: First occurrence of hospitalized angioneurotic oedema, pneumonia, gastroenteritis, failure to thrive, convulsions/seizures, acute interstitial nephritis and thrombocytopenia | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ron M.C. Herings, PhD, Principal Investigator — PHARMO Institute for Drug Outcome Research, Utrecht, The Netherlands; Leanne M.A. Houweling, MSc, Principal Investigator — PHARMO Institute for Drug Outcome Research, Utrecht, The Netherlands
Locations (1):
- Reserach Site, Utrecht, Netherlands

REFERENCES:
- [Derived] Houben E, Johansson S, Nagy P, Penning-van Beest FJA, Kuipers EJ, Herings RMC. Observational cohort study: safety outcomes in children using proton pump inhibitors or histamine-2 receptor antagonists. Curr Med Res Opin. 2018 Apr;34(4):577-583. doi: 10.1080/03007995.2017.1407302. Epub 2017 Nov 24. PMID 29149805
- [Derived] Ruigomez A, Kool-Houweling LMA, Garcia Rodriguez LA, Penning-van Beest FJA, Herings RMC. Characteristics of children and adolescents first prescribed proton pump inhibitors or histamine-2-receptor antagonists: an observational cohort study. Curr Med Res Opin. 2017 Dec;33(12):2251-2259. doi: 10.1080/03007995.2017.1336083. Epub 2017 Jun 9. PMID 28562108
- See also: D9612N00016 Children Study report synopsis Final redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=673&filename=D9612N00016%20Children%20Study%20report%20synopsis%20Final%20redacted.pdf